CLINICAL TRIAL: NCT06743477
Title: Clinical Study Protocol for Ultra-transplantation for the Treatment of Eastern Mediterranean Major
Brief Title: A Clinical Study of Ultra-transplantation for the Treatment of Major Thalassemia Scheme
Acronym: UTTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hu Peng (Other)
Responsible Party: Sponsor-Investigator, Hu Peng, Deputy Chief Physician, The First People's Hospital of Yunnan
Organization: The First People's Hospital of Yunnan (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KHLL2024-KY216; Hu Peng (Other: The First People's Hospital of Yunnan Province)
Record Dates: First submitted 2024-11-24; First posted 2024-12-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supergraft (Experimental): Hypertransplantation is an innovative treatment plan of Professor Ai Huisheng's team, which uses hematopoietic stem cell transplantation from healthy donors who are haplotype compatible with the patient, and observes the patient's cell reinfusion response, hematopoietic reconstitution, hemoglobin level and blood transfusion, thalassemia clonal clearance, immune reconstitution, endocrine function recovery, gastrointestinal function recovery, as well as the incidence of graft-versus-host disease, infection and other complications after transplantation.
  Interventions: Other: Supergraft

INTERVENTIONS:
Other: Supergraft — This study is a prospective, single-center, single-arm clinical study, and it is planned to include 3-5 patients with Eastern Mediterranean major who have no HSCT indication and cannot undergo Eastern Mediterranean gene therapy. The diagnosis of Eastern Mediterranean major was determined by the genotype of Eastern Mediterranean and the clinical manifestations of patients, and patients who met the inclusion criteria were screened and enrolled and received super transplant therapy.

SUMMARY:
Yunnan is a high-incidence area of Eastern Mediterranean (thalassemia) in China, and the treatment cost of thalassemia patients is high, hematopoietic stem cell transplantation (HSCT) is the only means to cure thalassemia, but there are problems in donor screening and the risk of complications. Professor Ai Huisheng's team proposed a new concept of hypertransplantation, which does not require pretreatment and has no risk of GVHD, and animal experiments have shown good efficacy. Under the guidance of Professor Ai, the center plans to carry out clinical research on hypertransplantation and explore safe and effective new therapies for thalassemia.

DETAILED DESCRIPTION:
Thalassemia (thalassemia, referred to as "ground poverty"), the incidence rate of birth defects in the third place, is a major public health problem worldwide. Yunnan is located in the subtropical region, adjacent to Southeast Asia, and is one of the high incidence areas of hemoglobinopathy in China. Its carrier rates of abnormal hemoglobinopathy and thalassemia are high, with obvious uniqueness and diversity. The detection rate of thalassemia carriers in the province is about 10.71%, while Dehong Prefecture, Xishuangbanna Prefecture, and Wenshan Prefecture are even higher at over 20.1%. Based on this, it is estimated that the number of patients with moderate to severe thalassemia in Yunnan is about 97000. The common treatments for patients with thalassemia include blood transfusion and hematopoietic stem cell transplantation. The cost of hematopoietic stem cell transplantation for each patient with thalassemia is approximately 250000 to 300000 yuan. The economic burden of blood transfusion treatment for children with thalassemia is greater and increases with age. A 1-year-old child with thalassemia requires approximately 20000 milliliters of blood per year, with an annual treatment cost of about 100000 yuan; To ensure the patient's survival at the age of 40, a total of approximately 4 million RMB is required. Such high treatment costs are difficult for ordinary families to afford. Hematopoietic stem cell transplantation (HSCT) is the only definitive treatment for thalassemia, and the development of clinical and basic research on gene therapy has led to a success rate of around 70%. HSCT and gene therapy both require pre-treatment with radiation, chemotherapy, and immunosuppression. The complications of HSCT include multi organ dysfunction caused by pre-treatment drugs, poor stem cell implantation, acute and chronic GVHD, some special complications (such as capillary leak syndrome (CLS), sinusoidal occlusion syndrome (SOS), interstitial pneumonia, thrombotic microvascular disease (TMA), post transplant lymphoproliferative disease (PTLD), hemorrhagic cystitis, central nervous system complications, etc.), which seriously affect the prognosis and quality of life of patients and cause varying degrees of damage to the reproductive development of children. HSCT supplier screening is also an urgent issue that needs to be addressed. The 5-year survival rate of MSD donor transplantation is 95-97%, but the sibling matching rate is 25%; The 5-year survival rate of MUD plants is 90-95%. Our province is a multi-ethnic mixed population, and the HLA polymorphism is significantly different from other Han ethnic populations. The success rate of non blood related matching is very low; The 5-year survival rate of haplotype donor transplantation is 80-87%, and the incidence of complications is significantly increased. Long term blood transfusion, high bone marrow load hematopoiesis, and irregular iron removal treatment are common among patients with thalassemia in China. The incidence of liver iron abnormalities is 89%, and the incidence increases with age. Long term anemia leading to heart damage, liver iron deposition, and other factors significantly reduces the success rate and long-term productivity of HSCT in critically ill thalassemia patients aged ≥ 7 years compared to patients aged<7 years, and most patients over 19 years old miss the opportunity for HSCT. Our province has long been in a backward state of economic and social development. Due to non-standard treatment of thalassemia and a shortage of MUD donors, there are many severe thalassemia patients who do not have the conditions for transplantation. Therefore, finding safer, more effective, and low-cost treatment strategies for severe thalassemia patients without transplantation conditions is a key challenge for the prevention and treatment of thalassemia in our province and even in the whole country and the world.

As is well known, Professor Ai Huisheng's team was the first to carry out non myeloablative transplantation (NST) in Asia and China in the late 1990s, and led the Chinese Non myeloablative Transplantation Collaboration Group. Afterwards, in 2011, they independently conducted micro transplantation and organized and led the International Micro Transplantation Interest Research Group internationally. Micro transplantation is simple, effective, and very safe, with almost no GVHD; Micro transplantation has received widespread support and replication applications both domestically and internationally. On this basis, Professor Ai's team has gone through more than ten years of research and exploration, and has innovatively proposed and developed new theories and models for super transplantation. Hypertransplantation does not require any pre-treatment of the recipient, nor does it use any cytotoxic drugs, radiotherapy, chemotherapy, or immunosuppressants. Through mutual immune reactions between the donor and recipient, a completely stable donor implantation (FDC) is ultimately formed. The results of animal experiments showed that even without any GVHD prevention, successful transplant recipients did not develop GVHD. At present, Professor Ai's team has conducted pioneering research on super transplantation, including animal experiments using C57BL/6 male mice as donor mice and CB6F1 β 654 female mice as transplant recipients; Experimental study on super transplantation of H2 haploidentical leukemia mice and thalassemia recipients. Especially in the super transplantation treatment of mice with thalassemia, all mice were not subjected to any GVHD pretreatment or GVHD prevention. However, all mice were able to form stable complete donor implants, and the thalassemia gene was reduced to an extremely low level close to zero; Hemoglobin, red blood cell count, white blood cell count, and platelet count all returned to normal levels in mice; Significant recovery of peripheral blood lymphocytes and thymus, and completion of immune reconstruction; Moreover, no acute or chronic GVHD was observed in the mice. In addition, the reproductive gland structure of female mice in the super transplantation group was intact after transplantation, and they were able to conceive, give birth, and breastfeed offspring normally. The good results of super transplantation in animal experiments of thalassemia are a major breakthrough in the treatment of thalassemia, and also lay a very good foundation for our upcoming clinical research on super transplantation of thalassemia.

Our center is the earliest unit in our province to carry out HSCT treatment for hematological diseases. The HSCT technology level is leading in the province, and we have solid clinical application conditions and foundations. We are willing to accept and adopt the new concept and treatment of super transplantation from Professor Ai Huisheng's team. Under Professor Ai's guidance and assistance, we will conduct clinical research on super transplantation for the treatment of severe thalassemia, verify its "safety and effectiveness", cure patients, and promote the continuous development of science, creating a safe and effective new treatment model for severe thalassemia without pre-treatment, reproductive damage, and post transplant complications.

ELIGIBILITY:
Patient inclusion criteria :

* Diagnosed with severe Mediterranean anemia, with no restrictions on alpha and beta types;
* Age between 7-12 years old, male or female not limited; Weight<40kg
* The patient has or does not have HLA matched or semi matched donors, but unconditionally transplants or refuses to undergo blood stem cell transplantation treatment; And patients who unconditionally or refuse to undergo gene therapy for thalassemia;
* There are HLA matched or mismatched donors who meet the donor criteria through physical examination;
* The patient and their family agree to receive super transplantation treatment and sign a written informed consent form before the transplantation trial.

  （2） Exclusion criteria for patients:
* Psychiatric patients;
* Participants in clinical trials of other drugs within the past month;
* There are no suitable HLA mismatched donors available.
* Other researchers have determined that they are not suitable to participate in this study.

  （3） Supplier screening criteria:
* HLA typing matches the patient's haplotype
* KIR configuration
* NIMA
* DSA negative
* Routine physical examination
* Genetic screening for carriers of thalassemia, mild or no carriers of thalassemia
* Sign the informed consent form.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-08-29 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Donor cell implantation rate | 3 months after transplantation
  Using polymerase chain reaction (PCR) to amplify short tandem repeat sequences Monitor the chimerism status of the donor and recipient to quantitatively evaluate the implantation rate of donor cells. Specifically, we will determine the percentage of donor cells and evaluate the implantation rate by comparing the DNA sequence differences between donor and recipient cells before and after transplantation.

SECONDARY OUTCOMES:
carriers of the Mediterranean anemia gene | one year
  Determine the status of carriers of Mediterranean anemia genes through gene sequencing technology. We will use specific molecular genetic methods, such as PCR and DNA sequencing, to identify and confirm specific mutations in the Mediterranean anemia gene.

OTHER OUTCOMES:
evaluation of growth and development | one year
  We will use standard assessment tools for children's growth and development, such as：
  Height Assessment:
  Outcome measure: Height in meters (m). Description: Monitor children's height growth and compare with standard data for children of the same age.
  weight assessment: Outcome measure: Body weight in kilograms. Description: Monitor children's weight gain and compare with standard data for children of the same age.
  Head circumference assessment:
  Outcome measure: Head circumference in centimeters (cm). Description: Monitor the growth of head circumference in children and compare it with standard data for children of the same age.
  Body mass index (BMI) assessment (if combined height and weight are required):
  Outcome measures: Body mass index (BMI) was measured in kg/m^2. Description: BMI values are obtained by calculating the weight (kg) divided by the square of height (m) to assess the proportion of a child's weight relative to height.

CONTACTS AND LOCATIONS:
Overall Officials: Yang T Yang, master, Principal Investigator — The First People's Hospital of Yunnan
Locations (1):
- Yunnan First People's Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing program aims to enhance research transparency and reproducibility, ensuring the validity of research results. We plan to release the raw data, including metadata and case record table data, within 6 months after the end of the trial. The data will be open for query through the clinical trial public management platform or directly provided to researchers. We use an electronic data collection and management system (EDC) for data collection and management to ensure data quality. During the sharing process, we will strictly adhere to privacy protection principles and safeguard individual privacy. This move is expected to promote scientific openness and information exchange, and deepen the value of clinical trial research. Despite the challenges, we are committed to promoting data sharing to enhance the credibility of medical research.
Supporting Information: Study Protocol, ICF
Time Frame: within 6 months after the end of the trial
Access Criteria: The IPD and supporting information will be accessible to researchers, academics, and the public with a legitimate interest in the study. They will be able to access the raw data, including metadata and case record form data, which are essential components of the study. Access to this data will be facilitated through a clinical trial public management platform, where the IPD will be openly available for query. Additionally, interested parties can directly contact the researchers to request access to the data. This approach ensures that the data is not only available to those within the scientific community but also to the general public, promoting transparency and broadening the impact of the research findings.

DOCUMENTS (2):
  • Study Protocol (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT06743477/Prot_000.pdf
  • Informed Consent Form (2024-12-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT06743477/ICF_001.pdf